CLINICAL TRIAL: NCT02843776
Title: Requests for Euthanasia and Assisted Suicide : Epidemiological Study Conducted as Part of the Establishment of a Structured Network
Brief Title: Requests for Euthanasia and Assisted Suicide
Acronym: EPIDESA2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Centre Hospitalier Pontarlier (Unknown); Centre Hospitalier de Haute Saône (Unknown); Centre Hospitalier du Val de Saône (Unknown); Centre Hospitalier Louis Pasteur (Unknown); Centre Hospitalier Champagnole (Unknown); Centre Hospitalier Lons le Saunier (Unknown); Centre Hospitalier Saint Claude (Unknown); Centre Hospitalier Belfort Montbéliard (Unknown); Centre Hospitalier Beaune (Unknown); Centre Hospitalier Chatillon Montbard (Unknown); Centre Hospitalier de l'Agglomération de Nevers (Other); Centre Hospitalier William Morey - Chalon sur Saône (Other); Centre Hospitalier Macon (Other); Centre Hospitalier de Monceau les Mines (Unknown); Centre Hospitalier Paray le Monial (Unknown); Centre Hospitalier Sens (Unknown); Centre Hospitalier Auxerre (Unknown); Centre Hospitalier Tonnerre (Unknown); Centre Hospitalier Joigny (Unknown); Réseau Opale (Unknown); Réseau Départemental de Soins Palliatifs de la Nièvre (Unknown); Groupement des Professionnels de Santé du Pays Beaunois (Unknown); Réseau ARESPA (Unknown); Réseau Pléiade (Unknown)
Responsible Party: Sponsor
Other Study IDs: EPIDESA2
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2016-07

CONDITIONS: Suicide, Assisted
Keywords: Palliative Care; Euthanasia; Epidemiologic Studies
MeSH Terms: conditions — Suicide, Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Questionnaires completion

SUMMARY:
The study epiDESA2 identifies all explicit requests for euthanasia or assisted suicide expressed by the person him/herself, regardless of which professional is asked and regardless of where the request is made (primary care, health institutions, medico-social institutions including nursing home care or at home) in the Burgundy-Franche-Comté region during six months.

ELIGIBILITY:
Inclusion Criteria:

Any adult :

* Living at home, or in medico-social institutions or hospitalized in primary care or health institutions of Burgundy-Franche-Comté,
* At the end of life due to advanced stage disease or a major change in the state of health of an elderly person,
* Who expressed an explicit request for euthanasia or assisted suicide,
* Who expressed their no objection to the collection of their datas,
* Who are covered by the French social security system.

Exclusion Criteria:

* They are underage
* The request was expressed by another person
* The request is not an explicit request
* The request appears in the context of a situation other than illness or a general change in state of health
* The patient is mentally confused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study epiDESA2 identifies all explicit requests for euthanasia or assisted suicide expressed by the person him/herself regardless of where the request is made (primary care, health institutions, medico-social institutions including EHPADs or at home) in the regions of Burgundy-Franche-Comté during six months.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Census of requests for euthanasia or assisted suicide in Burgundy-Franche-Comté | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No